CLINICAL TRIAL: NCT07057505
Title: Assesment of Pain, Foot Function, and Ultrasonographic Evaluation of Plantar Fascia Thickness in Patients Treated With Local Corticosteroid Injection for Plantar Fasciitis
Brief Title: Pain and Fascia Thickness After Steroid Injection in Plantar Fasciitis
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, mehmet tekne, Resident Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: 2025-41
Record Dates: First submitted 2025-07-07; First posted 2025-07-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; plantar fascia thickness; ultrasonographic evaluation; injection
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Plantar Fasciitis Patients with Corticosteroid Injection: The study cohort consists of patients clinically diagnosed with plantar fasciitis who have received local corticosteroid injections as part of their treatment. These patients were selected based on clinical criteria for plantar fasciitis and have undergone at least one ultrasound-guided corticosteroid injection targeting the affected plantar fascia.

SUMMARY:
The aim of this study is to evaluate the effects of local corticosteroid injection on pain, foot function index, and plantar fascia thickness in patients clinically diagnosed with plantar fasciitis, and to determine whether local corticosteroid injection is an appropriate treatment option for plantar fasciitis. For this purpose, the study plans to assess plantar fascia thickness using ultrasonography, evaluate pain using the Visual Analog Scale (VAS), and investigate the impact on daily living activities in patients who have been clinically diagnosed with plantar fasciitis and treated with local corticosteroid injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were clinically diagnosed with plantar fasciitis and received corticosteroid injections

Exclusion Criteria:

* Pregnancy
* Patients who have had more than one corticosteroid injection in the last 6 months
* Patients with systemic inflammatory diseases
* Patients who have previously undergone surgery in the heel area
* Patients with a history of local trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 33 patients who volunteered to participate in the study and applied to the Physical Medicine and Rehabilitation Clinic of the SBÜ Istanbul Physical Therapy and Rehabilitation Education and Research Hospital and were diagnosed with plantar fasciitis clinically and received local corticosteroid injections will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Plantar fascia thickness | The thickness measurement will be evaluated immediately after the injection and 1 month after the injection.
  Plantar fascia thickness measured by ultrasound
Pain score | Pain will be assessed with a visual analog scale immediately after injection and 1 month later
  Pain score assessed with a visual analog scale between 0 and 100

SECONDARY OUTCOMES:
Foot functions | Foot functions will be assessed immediately after injection and 1 month after injection with the foot function index.
  Foot functions will be assessed immediately after injection and 1 month after injection with the foot function index.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Tekne, Resident Doctor, Principal Investigator — Istanbul physical therapy rehabilitation training and research hospital; Nurdan Paker, Professor Doctor, Study Director — Istanbul physical therapy rehabilitation training and research hospital
Locations (1):
- Istanbul physical therapy rehabilitation training and research hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ''Yalıman A, Şen Eİ, Eskiyurt N, Budiman-Mak E. Ayak Fonksiyon İndeksi'nin Plantar Fasiitli Hastalarda Türkçe'ye Çeviri ve Adaptasyonu. Türk Fiz Tıp Rehab Derg 2014;60:212-22''
- [Background] Aggarwal P, Jirankali V, Garg SK. Evaluation of plantar fascia using high-resolution ultrasonography in clinically diagnosed cases of plantar fasciitis. Pol J Radiol. 2020 Jul 24;85:e375-e380. doi: 10.5114/pjr.2020.97955. eCollection 2020. PMID 32817771
- [Background] McMillan AM, Landorf KB, Gilheany MF, Bird AR, Morrow AD, Menz HB. Ultrasound guided corticosteroid injection for plantar fasciitis: randomised controlled trial. BMJ. 2012 May 22;344:e3260. doi: 10.1136/bmj.e3260. PMID 22619193